CLINICAL TRIAL: NCT05722717
Title: Genetic Risk Factors for Multi-system Inflammatory Syndrome in Children and Pediatric Post COVID Condition
Acronym: GRIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, epbuddingh, Dr. E.P. Buddingh, Leiden University Medical Center
Other Study IDs: NL80853.058.22
Record Dates: First submitted 2023-02-09; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: COVID-19; Post-Acute COVID-19; Post-Acute COVID19 Syndrome; Multi-System Inflammatory Syndrome in Children; Pediatric Inflammatory Multisystem Syndrome; Post COVID-19 Condition; Post-COVID-19 Syndrome
Keywords: COVID-19; Post-COVID Condition; MIS-C; PIMS-TS
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MIS-C: Children with a history of MIS-C: as defined according to WHO criteria, who were 0-18 at the time of MIS-C.
  Interventions: Genetic: Saliva collection at home
- Post COVID-Condition: Children with post-COVID condition who were 0-18 at the time of SARS-CoV-2 infection: as defined according to the WHO case definition.
  Interventions: Genetic: Saliva collection at home
- Control: 'Exposed' control group: children with a history of proven SARS-CoV-2 infection (RT-PCR, antigen test or serology positive) who were 0-18 at the time of SARS-CoV-2 infection.
  Interventions: Genetic: Saliva collection at home

INTERVENTIONS:
Genetic: Saliva collection at home — Children (with help of their parents) collect their saliva with a saliva collection kit which they send to our research center.

SUMMARY:
We will perform Whole Exome Sequencing on DNA from saliva. We will include: Children with a history of MIS-C; children with post-COVID condition; and controls in order to identify rare, high impact genetic variants in immunological genes and pathways in children with a history of MIS-C or pediatric post-COVID condition.

DETAILED DESCRIPTION:
Rationale:

Following infection with SARS-CoV-2, some children develop the potentially life-threatening disease Multi-System Inflammatory Syndrome in Children (MIS-C) and some children develop post-COVID condition (formerly 'long COVID'). It is unknown why some children develop severe or prolonged symptoms after SARS-CoV-2 infection, while most children have asymptomatic or mild disease. We hypothesize that rare variants in genes associated with the immune system predispose children to develop MIS-C or post-COVID condition after infection with SARS-CoV-2.

Objective:

Primary objective: To identify rare, high impact genetic variants in immunological genes and pathways in children with a history of MIS-C or pediatric post-COVID condition.

Secondary objectives: To analyze the clinical characteristics and long-term effects of pediatric COVID-19 and MIS-C. To characterize the functional and clinical impact of genetic variants in MIS-C and post-COVID condition and identify targets for therapy.

Study design:

We will do an observational study. We will perform Whole Exome Sequencing (WES) using Next Generation Sequencing (NGS) on DNA from blood or saliva. We will include: (1) MIS-C cases: Children with a history of MIS-C; (2) post-COVID condition cases: Children with post-COVID condition; and (3) Controls: SARS-CoV-2 exposed age-matched control group: children who were infected with SARS-CoV-2 but did not develop moderate to severe COVID-19, MIS-C or post-COVID condition.

Study population:

Children 0-19 years old with a history of MIS-C (n=100), post-COVID condition (n=100), or uncomplicated SARS-CoV-2 infection (n=200).

Main study parameters/endpoints:

1. To evaluate if some children with MIS-C or post-COVID condition have an inborn error of immunity by determining the presence of pathogenic or likely pathogenic variants in immunological genes
2. To evaluate if a larger proportion of cases with MIS-C or post-COVID condition have rare and presumably deleterious variants in immunological genes than children with an asymptomatic or mild infection

ELIGIBILITY:
Inclusion Criteria:

1. Children (<19 years) with a history of MIS-C: as defined according to WHO criteria.
2. Children (<19 years) with post-COVID condition: as defined according to the WHO case definition. This includes a history of probable or confirmed prior SARS-CoV-2 infection, with signs and symptoms (including fatigue, shortness of breath, cognitive dysfunction) that are present after 12 weeks, last at least 2 months, have an impact on daily functioning and are not explained by an alternative diagnosis.
3. 'Exposed' control group: children (<19 years of age): a history of proven SARS-CoV-2 infection (RT-PCR, antigen test or serology positive). If the child has been vaccinated against SARS-CoV-2, the first documented infection must have been prior to the vaccination.

Exclusion Criteria:

1. No informed consent
2. Group 1 (MIS-C): no specific exclusion criteria
3. Group 2 (post-COVID condition): other plausible cause of symptoms AND/OR a history compatible with chronic fatigue syndrome prior to infection with SARS-CoV-2.

   Children with a history of MIS-C who suffer prolonged signs and symptoms will be included in the MIS-C group.
4. Group 3 ('exposed' control group): MIS-C or post-COVID condition; AND/OR Moderate or severe course of COVID-19, as defined in the COPP-study (N20.043) (need for supplemental oxygen and/or intensive care admission because of COVID-19 and/or death) AND/OR first degree relative with long COVID or MIS-C.

Ages: 0 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with a history of MIS-C or Post-COVID Condition and children with a known SARS-CoV-2 infection without severe disease course.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Quantity and quality of genetic variants in immunological genes between study groups. | 2 year
  We want to quantify how many immunogenic variants are found between the groups and identify which variants/genes these are.

SECONDARY OUTCOMES:
Correlate genetic findings with clinical characteristics | 2 year
  We want to connect the data found during genetic testing with multiple clinical characteristics already collected in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Emmeline P Buddingh, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided